CLINICAL TRIAL: NCT02401672
Title: Developing rTMS as a Potential Treatment for Nicotine Addiction
Brief Title: Repetitive Transcranial Magnetic Stimulation (rTMS) for Nicotine Addiction
Acronym: rTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Xingbao Li, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: pro00032313
Record Dates: First submitted 2015-03-16; First posted 2015-03-30 (Estimated); Results first posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-08

CONDITIONS: Nicotine Dependence
Keywords: TMS; nicotine dependence; smoking cessation
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active TMS (Active Comparator): Repetitive TMS pulse stimulation
  Interventions: Device: Transcranial magnetic stimulation
- Sham TMS (Sham Comparator): The sham TMS system will be connected to an electrical generator on a 9 V battery and electrodes will be placed over the prefrontal cortex. The regulator is triggered by the TMS machine to allow brief, microsecond, pulses of the electrical current through to the skin on the subjects' forehead. Electrical stimulation will be triggered by the TMS machine to correspond to the sham TMS pulses.
  Interventions: Device: Transcranial magnetic stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation — Transcranial magnetic stimulation (TMS) is a noninvasive (and relatively painless) brain stimulation technology that can focally stimulate the brain of an awake individual. A localized pulsed magnetic field transmitted through a TMS coil is able to focally stimulate the cortex by depolarizing superficial neurons inducing electrical currents in the brain. If TMS pulses are delivered repetitively and rhythmically, the process is called repetitive TMS (rTMS).

SUMMARY:
Cigarette smoking remains a significant public health concern. A magnetic field applied to the outside of the skull can produce electrical activity in the brain without significant pain or the need for anesthesia. Sessions of magnetic stimulation or superficial stimulation that does not reach the brain will be used to determine if magnetic stimulation can reduce cue-induced craving and cigarettes consumption in adult nicotine-dependent cigarette smokers. This project may lead to a new therapy for smoking cessation.

DETAILED DESCRIPTION:
Cigarette smoking causes significant morbidity and mortality in the United States. Smoking cessation is difficult, with the average smoker attempting to quit five times before permanent success. Moreover, the majority of smoking quit attempts result in relapse. Brain stimulation for smoke cessation is an exciting new area that builds on advancing neuroscience knowledge concerning the functional neurocircuitry of addiction. Cortical stimulation can now be performed non-invasively by transcranial magnetic stimulation (TMS). A few studies have shown that TMS can reduce cue-elicited craving in smokers. Previous research by our group has shown that a single session of 15 minutes high frequency (10 Hz) repetitive TMS (rTMS) at 100% motor threshold over the left dorsal lateral prefrontal cortex (an area that is likely involved in inhibiting craving) can reduce cue-induced craving compared to sham TMS. However, methodological concerns surrounding these preliminary findings limit definitive conclusions about the effectiveness of TMS over a longer period of time. This R21 proposal will integrate more rigorous experimental conditions, a true double-blind methodology, MRI guided stimulation site and a longer-term follow-up assessment. Using rigorous double-masked methods and MRI guided stimulation site, we propose that using active rTMS or sham rTMS, to determine whether 10 sessions over a two week period consisting of 15 minute high frequency rTMS can reduce cue-induced craving and cigarette consumption for cigarette smokers. The project will also optimize rational rTMS parameters to make TMS to an efficacious treatment for nicotine dependence. In the two years of project, we plan to recruit 42 treatment-seeking nicotine-dependent cigarette smokers, both males and females of all ethnic and racial groups between the ages of 18 and 60 to participate in the study. The 42 participants will be randomly assigned to receive active prefrontal TMS or sham prefrontal TMS. The data from this R21 will provide the information needed for launching a definitive larger-scale investigation into potential clinical applications of TMS in smoke cessation. The results from this pilot will also likely supply substantial information about the utility of cortical stimulation for smoke cessation.

ELIGIBILITY:
Inclusion Criteria:

1. Be between the ages of 18 and 60 years old.
2. Smoke 10 or more cigarettes per day and have a carbon monoxide (CO) level > 10 ppm indicative of recent smoking.
3. Not received substance abuse treatment within the previous 30 days.
4. Meet criteria for nicotine dependence as determined by the FTND.
5. Be in stable mental and physical health.
6. If female, test non-pregnant and use adequate birth control.
7. No evidence of focal or diffuse brain lesion on MRI.
8. Be willing to provide informed consent.
9. Be able to comply with protocol requirements and likely to complete all study procedures.

Exclusion Criteria:

1. Current dependence, defined by DSM-V criteria, on any psychoactive substances other than nicotine or caffeine.
2. Contraindication to MRI (e.g., presence of metal in the skull, orbits or intracranial cavity, claustrophobia).
3. Contraindication to rTMS (history of neurological disorder or seizure, increased intracranial pressure, brain surgery, or head trauma with loss of consciousness for > 15 minutes, implanted electronic device, metal in the head, or pregnancy).
4. History of autoimmune, endocrine, viral, or vascular disorder affecting the brain.
5. History or MRI evidence of neurological disorder that would lead to local or diffuse brain lesions or significant physical impairment.
6. Unstable cardiac disease, uncontrolled hypertension, severe renal or liver insufficiency, or sleep apnea.
7. Life time history of major Axis I disorders such as: Bipolar Affective disorder (BPAD), Schizophrenia, Post-traumatic Stress disorder (PTSD) or Dementia or Major Depression.
8. Self report of >21 standard alcohol drinks per week in any week in the 30 days prior to screening.
9. Other forms of nicotine delivery, such as nicotine patch, electronic cigarettes

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2014-05-14 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li X, Hartwell KJ, Owens M, Lematty T, Borckardt JJ, Hanlon CA, Brady KT, George MS. Repetitive transcranial magnetic stimulation of the dorsolateral prefrontal cortex reduces nicotine cue craving. Biol Psychiatry. 2013 Apr 15;73(8):714-20. doi: 10.1016/j.biopsych.2013.01.003. Epub 2013 Feb 26. PMID 23485014
- [Derived] Li X, Caulfield KA, Hartwell KJ, Henderson S, Brady KT, George MS. Reduced executive and reward connectivity is associated with smoking cessation response to repetitive transcranial magnetic stimulation: A double-blind, randomized, sham-controlled trial. Brain Imaging Behav. 2024 Feb;18(1):207-219. doi: 10.1007/s11682-023-00820-3. Epub 2023 Nov 23. PMID 37996557
- [Derived] Li X, Hartwell KJ, Henderson S, Badran BW, Brady KT, George MS. Two weeks of image-guided left dorsolateral prefrontal cortex repetitive transcranial magnetic stimulation improves smoking cessation: A double-blind, sham-controlled, randomized clinical trial. Brain Stimul. 2020 Sep-Oct;13(5):1271-1279. doi: 10.1016/j.brs.2020.06.007. Epub 2020 Jun 10. PMID 32534252

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Assessed for eligibility (n=327), Excluded 280, Not meeting inclusion criteria: 275, and declined to participate: 5, lost contact before screening visit: 5
Period: Overall Study
Arm/Group | Active TMS | Sham TMS
Started | 22 | 20
Completed | 21 | 17
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Population: This study is a randomized, double-blinded, sham-controlled trail. The active group has 2 more participants than the sham. However, this is acceptable for the small sample size trial. Especially, this is from randomized trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active TMS | Sham TMS | Total
Number analyzed (Participants) | 22 | 20 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] — the length of years started his/her birth date.
  years | 40.64 (10.36) | 43.75 (10.36) | 42.12 (10.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 10 | 9 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 19 | 19 | 38
  Race: African Americans | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 20 | 42
cigarettes per day [Mean (Standard Deviation); unit: cigarettes per day] | 18.2 (4.8) | 20.9 (10.2) | 19.5 (7.8)

OUTCOME MEASURES:

1. Primary Outcome: Nicotine Consumption: Number of Cigarettes Per Day
Description: Nicotine consumption: We use cigarette diary for participant to record number of cigarettes smoked per day.
Time Frame: 2 weeks of treatment
Population: two groups t test for percentage changed cigarettes per day: mixed model.
Measure: Mean (Standard Deviation); unit: the number of cigarette
Arm/Group | Active TMS | Sham TMS
Number analyzed (Participants) | 21 | 17
the number of cigarette | 11.60 (6.93) | 13.73 (9.18)
Statistical Analysis 1: Comparison: Active TMS vs Sham TMS; Test type: Superiority; p = 0.05, Mixed Models Analysis

2. Primary Outcome: Percentage of Change of Cigarettes Per Day
Description: percentage of change of cigarettes per day =100* ( cigarettes smoked per day at baseline - cigarettes smoked per day at the end of treatment) / cigarettes smoked per day at baseline
Time Frame: 2 weeks
Population: We compared active group to sham group in the percentage of reduction in cigarettes smoked per day.
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Active TMS | Sham TMS
Number analyzed (Participants) | 21 | 17
% change | 62.93 (10.74) | 38.43 (10.63)
Statistical Analysis 1: Comparison: Active TMS vs Sham TMS; Test type: Superiority; p = 0.05, t-test, 2 sided

3. Secondary Outcome: Average Nicotine Craving as Assessed by the Questionnaire of Smoking Urges-Brief
Description: The Brief Questionnaire of Smoking Urges (QSU-Brief) consists of 10 statements about the respondent's feelings and thoughts about his or her desire to smoke cigarettes as he or she is completing the questionnaire. A higher number represents a stronger smoking urges. A lower score represents a weaker smoking urges. The lowest score is 10. The highest score is 70.
Time Frame: 2 weeks of treatment
Population: Weekly ratings for mixed model repeated measures. We reported the group means which includes 5 points each group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active TMS | Sham TMS
Number analyzed (Participants) | 21 | 17
score on a scale | 25.01 (14.45) | 29.93 (13.12)
Statistical Analysis 1: Comparison: Active TMS vs Sham TMS; Test type: Superiority; p = 0.05, Mixed Models Analysis

4. Secondary Outcome: The Number of Participants Quitting on the Target Quit Date
Description: Quitting smoking on the target quit date.
Time Frame: 2 weeks of treatment
Population: Quitting at target quit date.
Measure: Number; unit: participants
Arm/Group | Active TMS | Sham TMS
Number analyzed (Participants) | 21 | 17
participants | 5 | 0
Statistical Analysis 1: Comparison: Active TMS vs Sham TMS; Test type: Superiority; p = 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: Two weeks
Description: When the active TMS treatment started, the participant could not be tolerable for the stimulation. The participant dropped out the study.
  We asked for any side effects during the treatment course. E.g. Headache, discomfort, unpleasant or scalp pain.
Arm/Group | Active TMS | Sham TMS
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/17
Other Adverse Events (participants affected / at risk) | 14/21 | 8/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active TMS (N=21) | Sham TMS (N=17)
headache (Nervous system disorders) | 14 (14) | 8 (8) — Headache, discomfort , unpleasant or scalp pain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-21): https://cdn.clinicaltrials.gov/large-docs/72/NCT02401672/Prot_SAP_000.pdf